CLINICAL TRIAL: NCT04868734
Title: Development of a Superficial Supportive Psychotherapy Model and Its Effect on Acute Coronary Syndrome Patients Psycho-Neuro-Endocrine Studies
Brief Title: Superficial Supportive Psychotherapy Model and Its Effect on Acute Coronary Syndrome Psycho-Neuro-Endocrine Studies
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Hamzah Shatri, Principle Investigator, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 20-11-1478
Record Dates: First submitted 2021-04-20; First posted 2021-05-03 (Actual); Last update posted 2022-03-15 (Actual); Status verified 2022-03

CONDITIONS: Psychosomatic Disorder
Keywords: Psychotherapy Supportive
MeSH Terms: conditions — Psychophysiologic Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supportive Psychotherapy (Experimental): Supportive Psychotherapy do to subjects
  Interventions: Behavioral: Supportive Psychotherapy
- Casual Treatment (No Intervention): Do Casual Intervention

INTERVENTIONS:
Behavioral: Supportive Psychotherapy — Supportive Psychotherapy give to patient with Acute Coronary Syndrome
  Arms: Supportive Psychotherapy

SUMMARY:
Hypothesis

1. The supportive psychotherapy model can be structured and developed for the non-pharmacologic therapy of acute coroner syndrome patients in intensive cardiac care unit
2. The development of the supportive psychotherapy model can provide an improvement in psychological function in the form of a reduction in symptoms of anxiety, depression, and an improvement in the quality of life of acute coroner syndrome patients during treatment at intensive cardiac care unit.
3. Psycho-patho-mechanization of supportive psychotherapy model development in the improvement of psychosomatic function of acute coroner syndrome patients by assessing the improvement of serotonin, cortisol, and immunoglobulin-A levels, and,
4. Development of the supportive psychotherapy model can provide improvement in somatic function in the form of decreased complications such as arrhythmias, pericarditis, chronic heart failure, shock and death of acute coronary syndrome patients during treatment.
5. Psychosomatic improvements, namely anxiety, depression, and cardiac complications associated with levels of serotonin, cortisol, immunoglobulin-A and heart rate variability.

Research objectives 1.1 General Objectives: To develop non-pharmacologic psychotherapy as part of holistic therapy for acute coronary syndrome patients during their treatment at intensive cardiac care unit.

1.2 Specific Objectives:

1. Develop a structured supportive psychotherapy model
2. Proving the role of supportive psychotherapy in the improvement of psychological symptoms of anxiety, depression and quality of life in acute coronary syndrome patients during treatment.
3. Proving the psycho-patho-mechanism intervention of the supportive psychotherapy model in improving psychosomatic function through the Hypothalamus-Pituitary-Adrenal pathway, namely by assessing the improvement in levels of serotonin, cortisol, immunoglobulin-A and heart rate variability
4. Proving the role of supportive psychotherapy in the improvement of somatic symptoms of cardiac complications such as arrhythmias, pericarditis, chronic heart failure, shock and death in acute coronary syndrome patients during treatment.
5. To prove the supportive psychotherapy model in psychosomatic improvement, namely anxiety, depression, and cardiac complications associated with improvements in levels of serotonin, cortisol, immunoglobulin-A and heart rate variability.

DETAILED DESCRIPTION:
Introduction Acute coronary syndrome will have a high impact on who feels it. Psycho-neuro-immunological imbalance will occur before and after the attack. To date, there is no evidence regarding the role of supportive psychotherapy as a non-medical treatment in acute coronary syndromes. The study will also measure cortisol, immunoglobulin-A, serotonin, and heart rate variability for objective comparisons between intervention and usual cardiac care.

Method This research is an operational research with a mixed method research design, namely exploratory sequential method with qualitative method research that precedes quantitative methods. This research is divided into two stages, namely the qualitative research stage by developing a model of supportive psychotherapy, followed by the stage of applying the model to clinical trials of acute coronary syndrome patients during treatment at intensive cardiac care unit.

Result Total subject is 80 subject. All will collect blood and saliva sample, heart rate variability. One arm will do intervention (supportive psychotherapy) and the others will do usual cardiac care.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years or older
2. Patients diagnosed with ACS by cardiologists and have received standard management with or without PCI.
3. The patient is willing to participate in the research

Exclusion Criteria:

1. ACS patients who had acute complications related to ACS upon admission before the study started, such as the presence of CHF, arrhythmias, pericarditis, cardiogenic shock or death.
2. Psychotic disorders (with delusions or psychosis)
3. Not willing to take part in research

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2021-04-07 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-12-30 (Actual)

PRIMARY OUTCOMES:
Changes Visual Analog Scale In Comfort Feeling after Superficial Supportive Psychotherapy Model on Acute Coronary Syndrome Patients | per subject will completed about 12 days. Supportive psychotherapy will do to intervention subject and all subject (wit and without intervention) will ask visual analog scale at day 1, day 5, and day 12.
  Visual Analog Scale measurement (in numeric scale from 0 to 10)

SECONDARY OUTCOMES:
Changes in blood serotonin levels after Superficial Supportive Psychotherapy Model on Acute Coronary Syndrome Patients | All subject will completed about 12 days. The blood sample will check at day 1, day 5, and day 12.
  Serotonin level measurement (ng/dL)
Changes in saliva cortisol levels after Superficial Supportive Psychotherapy Model on Acute Coronary Syndrome Patients | All subject will completed about 12 days. The saliva sample will check at day 1, day 5, and day 12.
  Cortisol level measurement (ng/dL)
Changes in saliva immunoglobulin-A levels after Superficial Supportive Psychotherapy Model on Acute Coronary Syndrome Patients | All subject will completed about 12 days. The saliva sample will check at day 1, day 5, and day 12.
  Immunoglobulin-A level measurement (ng/dL)

CONTACTS AND LOCATIONS:
Overall Officials: Hamzah Shatri, Principal Investigator — Indonesia University
Locations (1):
- dr Cipto Mangunkusumo Hospital, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided